CLINICAL TRIAL: NCT03218904
Title: Application of Novel Techniques to Devise Nutritional Therapies in Subjects with Glycogen Storage Disease Type I
Brief Title: Glycogen Storage Disease Breath Test Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Saudi Arabian Cultural Bureau, Ottawa (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: H16-03050
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Patient Compliance; Healthy
Keywords: Glucose Breath Test
MeSH Terms: conditions — Patient Compliance | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucose intake (Experimental): Experiment 1: study day 1- single oral dose of glucose study day 2- single oral dose of glucose with U-13C-glucose
  Interventions: Dietary Supplement: Glucose intake
- Carbohydrates intake (Experimental): Experiment 2: study day 1-single oral dose of uncooked cornstarch study day 2-single oral dose of Glycosade®
  Interventions: Dietary Supplement: Carbohydrates intake

INTERVENTIONS:
Dietary Supplement: Glucose intake — Experiment 1: study day1- single oral dose of glucose study day 2-single oral dose of glucose with U-13C-glucose
  Other Names: D-glucose (Thermo Scientific™ NERL™ Trutol™)
  Arms: Glucose intake
Dietary Supplement: Carbohydrates intake — Experiment 2:study day1- single oral dose of uncooked cornstarch study day 2- single oral dose of Glycosade®
  Other Names: Uncooked cornstarch; Glycosade®
  Arms: Carbohydrates intake

SUMMARY:
Glycogen storage disease type I (GSD I) caused by deficiency of glucose-6-phosphatase enzyme leading to build up of a complex sugar called glycogen in liver and low blood glucose level. Nutritional treatment involves supplying carbohydrates and uncooked cornstarch. Glycosade® (modified cornstarch) has shown promise in maintaining normal blood glucose level in GSD I. But the difficulty in nutritional treatment is determining the best type of carbohydrate to be given to avoid low blood glucose. Thus, there is a need to develop a simple test to examine glucose digestion and measure the utilization of different carbohydrates in GSD I and healthy controls.

DETAILED DESCRIPTION:
Purpose: Glycogen storage disease type I (GSD I), also known as Von Gierke disease is caused by deficiency of glucose-6-phosphatase (G6Pase) enzyme affecting 1:100,000 births worldwide. Therefore, deficiency of this enzyme results in accumulation of glycogen in liver and inadequate production of glucose leading to fasting hypoglycemia. Dietary treatment for GSD I is based on supplying complex carbohydrates with small frequent meals, and use of uncooked cornstarch (UCCS). Glycosade® (modified cornstarch) has shown promise in maintaining normal blood glucose concentrations in subjects with GSD I. However, the primary dilemma in the dietary treatment of GSD I is the choice of the exogenous carbohydrate sources to achieve a desirable metabolic control and prevent hypoglycemia. In addition, the previous studies were invasive, which required several blood samples, long study days (~10 h) and could not offer mechanistic details of glucose metabolism in subjects with GSD I. Thus, there is a need to develop a minimally-invasive method to examine glucose metabolism and measure the utilization of different carbohydrate sources directly in subjects with GSD I and healthy controls. This simple breath test will help individualize treatment and tailor carbohydrate supply in subjects with GSD I.

Hypothesis: 1) Investigators hypothesize that the oxidation of isotopic carbon dioxide (13CO2) from U-13C-glucose can be detected in expired air; and 13CO2 oxidation will be a sensitive measure to examine glucose oxidation/metabolism.

2) Investigators hypothesize that 13CO2 oxidation from Glycosade® will have lower peak enrichment (Cmax) compared to other carbohydrate source UCCS in patients with GSD I and healthy controls.

Justification: The difficulty in nutritional treatment of GSD I is determining the best type of carbohydrate to be given to avoid hypoglycaemia. Therefore glucose metabolism and the utilization of different carbohydrates need to be measured using minimally invasive test.

Objectives: 1) Our first objective is to establish the use of U-13C-glucose breath test (13C-GBT) and its oxidation to 13CO2 as a minimally-invasive technique to examine in vivo glucose oxidation in healthy controls.

2) Our second objective is to measure the utilization of different exogenous carbohydrate sources: UCCS and the extended release waxy maize cornstarch Glycosade® in healthy controls and patients with GSD I using a minimally invasive 13C-GBT.

Research Method: The project consists of two experiments.

Experiment 1 - Pilot Study to Establish the Use of U-13C-Glucose Breath Test (13C-GBT) in Healthy Controls A. Pre-study Day Protocol Written informed consent will be obtained from participants before participating in the study. All participants will be requested to fast overnight (~ 12 hours) and will be asked to come to the Clinical Research and Evaluation Unit for a preliminary assessment (pre-study day) to measure basic anthropometry (weight and height), body composition and resting energy expenditure (REE). Weight and height will be measured by using a digital scale and a stadiometer, respectively. REE will be measured by continuous, open-circuit indirect calorimetry (CareFusion Vmax Encore, VIASYS), which will be calibrated prior to use. Total energy expenditure (TEE) and basal metabolic rate (BMR) are associated to fat free mass (FFM); therefore body composition will be determined using bioelectrical impedance analysis (BIA) (Quantum IV RJL systems). BIA measures resistance, reactance and impedance by applying electrodes placed at the right wrist and right ankle. Three readings for resistance, reactance and impedance will be taken for each participant - then the mean of these readings will be used to determine FFM and fat mass (FM). FFM and FM will be calculated using the manufacturer's software system (RJL Systems, Body Composition Analysis V.2.1). A general questionnaire will be used during the pre-study day to give a clear idea about medical history, nutritional status, supplement intake and physical activity. Finally, 3-day dietary record sheets will be distributed to the participants to record food consumption for any two days during the week and one day on the weekend.

B. Two-Day Dietary Standardization During the two days prior to study, subjects will consume a balanced diet containing at least 150 g of carbohydrate. This diet consisted of everyday foods, however an outline will be given to subjects to ensure sufficiency based on foods commonly eaten.

C. Study day Protocol For pilot study, 10 healthy adults (19-35 y) will undergo 13C-GBT protocols in two separate study days as a proof-of-principle, once without oral isotope dose and once with oral isotope dose (U-13C-glucose), each study separated by ≥ 1 week. Thus, 10 healthy adults will be studied for a total of n = 20 studies. After obtaining informed consent from the subject, the subject will be enrolled in the study. The participant will arrive for the study day after fast (~4 h) to standardize measurements at the Clinical Research and Evaluation Unit (CREU) at British Columbia (BC) Children's Hospital. Basic anthropometric measurements (body weight and height) will be collected and a brief study day questionnaire will be administered to collect information on medical, diet and physical activity history. 2 Baseline breath samples will be collected to determine natural background 13C abundance. Subjects will receive on study day 1 glucose (75 g/day) dissolved in sterile water, study day 2 U-13C-glucose (75 mg/day) (99 atom% 13C enrichment, Cambridge Isotope Laboratories Inc., Andover, MA) with glucose (75 g/day) dissolved in sterile water.

Subjects will remain fasting and resting in CREU for the entire period of the study to eliminate variability in CO2 production. Breath samples in quadruplicates will be collected at 20,40,60,80,100,120,140,160,180, 200, 220 and 240 min after oral administration of glucose. During the study visit, the rate of carbon dioxide production (VCO2) will be measured for 20 minutes, two hours (120 minutes) after the oral glucose dose using an indirect calorimeter (Vmax Encore, Viasys Healthcare Inc. Yorba Linda, CA). Assessment of body composition will be performed using the Bioelectrical Impedance Analysis (BIA-Quantum IV, RJL Systems, MI). BIA calculated resistance, reactance and impedance by applying electrodes would be placed at the right wrist and ankle. Three readings for resistance, reactance and impedance will be taken for each subject then the mean of these readings will be used to determined fat free mass (FFM) and fat mass (FM). FFM and FM will be calculated using the manufacturer's software system (RJL Systems, Body Composition Analysis V.2.1). Finger-prick blood glucose samples will be assessed at the beginning and hourly until the end of the study day using glucometer (One Touch® Ultra®, LifeScan, Inc).

Sample Collection and Analysis: Breath samples will be collected using breath bags (single use collection bags, EasySampler System, QuinTron Instrument Company, Inc. Milwaukee, WI) in disposable glass Exetainer® tubes (Labco Limited, Buckinghamshire, UK) using a collection mechanism that permits removal of dead air space. The breath enrichment of 13CO2 will be measured using isotope ratio mass spectrometer (IRMS).

Statistical Analysis Subject characteristics will be expressed as the mean (SD). 13C-glucose oxidation as 13CO2 will be the primary outcome measured, as this best describes the whole body oxidation capacity for glucose. Area under the curve (AUC) for each subject's 13CO2 oxidation from t0 to t240, the time to reach maximum 13CO2 oxidation (tmax) and the maximum peak enrichment in 13CO2 oxidation (Cmax) will be calculated. A repeated-measures analysis using restricted maximum likelihood estimation will be used to get the estimated parameters with the MIXED procedure using SAS software (SAS/STAT; Version 9.2). A paired t-test will be used to compare the 13CO2 oxidation at each time point without and with U-13C-glucose. All values will be presented for individual subjects, and significance is set at P<0.05. Statistical analysis will be performed using GraphPad Prism 4.0 (GraphPad Software Inc, CA).

Experiment 2 - Minimally Invasive 13C-Glucose Breath Test to Measure the Utilization of Different Exogenous Carbohydrate Sources in Healthy Controls and Subjects with Glycogen Storage Disease Type I For initial set of studies, 10 healthy children (5-18 y) and 10 healthy adults (19-35 y) will undergo 13C-GBT four times. Then, 3 children and 5 adults with GSD I will be recruited in 4 separate study days from our Pediatric and Adult metabolic clinic at BC Children's and Vancouver General Hospital, respectively (if recruitment is a challenge, we plan to approach clinics across Canada). After fast (~ 4 h for healthy controls and 2 h for GSD I) subjects will receive on study day 1- UCCS (2 g/kg/day), study day 2- U-13C-glucose (75 mg for adults; 1.5 mg/kg for children) (99 atom% 13C enrichment, Cambridge Isotope Laboratories Inc., Andover, MA) with UCCS (2 g/kg/day), study day 3- the extended release waxy maize cornstarch Glycosade® (2 g/kg/day) (Vitaflo International Ltd, Liverpool, England), and on study day 4- U-13C-glucose (75 mg for adults; 1.5 mg/kg for children) with Glycosade® (2 g/kg/day) dissolved in sterile water. On each study day, breath samples will be collected every 20 min for 240 min. The rate of CO2 production will be measured at 120 min after oral dose using indirect calorimetry. Blood glucose will be measured using glucometer and finger-prick blood samples will be assessed at the beginning and hourly until the end of the study day. The percentage of test carbohydrates exhaled, as 13CO2 will be measured over a 4 h period.

Statistical Analysis Subject characteristics will be expressed as the mean (SD). 13C-glucose oxidation as 13CO2 will be the primary outcome measured, as this best describes the whole body oxidation capacity for glucose. Area under the curve (AUC) for each subject's 13CO2 oxidation from t0 to t240, the time to reach maximum 13CO2 oxidation (tmax) and the maximum peak enrichment in 13CO2 oxidation (Cmax) will be calculated for UCCS and Glycosade®. The values obtained from the carbohydrate sources will be compared by using a two-tailed paired t-test. Significance will be set at P<0.05.

Statistical analysis will be performed using GraphPad Prism 4.0 (GraphPad Software Inc, CA).

ELIGIBILITY:
Inclusion Criteria:

Experiment 1

* Healthy adults 19 - 35 years of age
* Adults who have no medical conditions
* Adults who currently free from any concurrent illness such as fever or cold

Experiment 2

Healthy Controls:

* Healthy children 5 - 18 years of age
* Healthy adults 19 - 35 years of age
* Children and adults who have no medical conditions
* Children and adults who currently free from any concurrent illness such as fever or cold

Subjects with GSD I:

* Children 5 - 18 years of age who are diagnosed with GSD I
* Adults 19 - 35 years of age who are diagnosed with GSD I
* Clinically stable children and adults with GSD I with no concurrent illness such as fever, cold, vomiting or diarrhea
* Children and adults with GSD I who have had the clinical decision made to start the extended release waxy maize cornstarch Glycosade®

Exclusion Criteria:

Experiment 1

* Healthy adults above age 35 years
* Adults who have a history of cardiovascular disease, liver or kidney disease, metabolic, pulmonary, gastrointestinal or endocrine disorder
* Healthy adults but are currently ill with a fever, cold, vomiting or diarrhea
* Healthy adults with claustrophobia
* Healthy adults currently smoking or consuming more than one drink containing alcohol each day
* Adults currently or recently taking medication or antibiotics

Experiment 2

Healthy Controls:

* Healthy children under age 5 years
* Healthy adults above age 35 years
* Children and adults who have a history of cardiovascular disease, liver or kidney disease, metabolic, pulmonary, gastrointestinal or endocrine disorder
* Healthy children and adults but are currently ill with a fever, cold, vomiting or diarrhea
* Healthy children and adults with claustrophobia
* Children and adults currently or recently taking medication or antibiotics
* Healthy adults currently smoking or consuming more than one drink containing alcohol each day

Subjects with GSD I:

* Children with GSD I under age 5 years
* Adults with GSD I above age 35 years
* Children and adults diagnosed with GSD I, but are currently ill with a fever, cold, vomiting or diarrhea
* Children and adults diagnosed with GSD I, but where the clinical decision has been made not to start on Glycosade®
* Children and adults with GSD I who have claustrophobia
* Children and adults with GSD I currently or recently taking medication or antibiotics
* Adults with GSD I currently smoking or consuming more than one drink containing alcohol each day

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Glucose oxidation | 4 hours
  Breath sample will be collected during the study to measure the rate of oxidation of 13C glucose

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with other researchers